CLINICAL TRIAL: NCT02290769
Title: Evaluation of the Cannulation Time During Primary ERCP With Short Guide Wire Rapid Exchange or With Long Guide Wire. Multicentre Prospective Randomized Trial
Brief Title: Time of Cannulation During Primary ERCP With Short Guide Wire Rapid Exchange or With Long Guide Wire
Acronym: RELG
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Hospital administrative problems
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 382 - 072014
Record Dates: First submitted 2014-10-27; First posted 2014-11-14 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Pancreatitis
Keywords: Guide wire cannulation ERCP; Time of cannulation; Rapid exchange guide wire; Guide wire
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short guide wire rapid exchange (Experimental): Use of short guide wire rapid exchange to guide the cannulation during primary ERCP
  Interventions: Device: Short guide wire rapid exchange
- Long guide wire (Active Comparator): Use of long wire to guide the cannulation during primary ERCP
  Interventions: Device: Long guide wire

INTERVENTIONS:
Device: Short guide wire rapid exchange — Use of short guide wire rapid exchange to guide the cannulation during primary ERCP
  Arms: Short guide wire rapid exchange
Device: Long guide wire — Use of long wire to guide the cannulation during primary ERCP
  Arms: Long guide wire

SUMMARY:
The aim of this study is to compare the cannulation time during primary wire guided ERCP (Endoscopic Retrograde Cholangio-Pancreatography) according to two different length of guide wire: long wire or short wire rapid exchange, artery by a prospective randomized trial.

DETAILED DESCRIPTION:
In primary Endoscopic Retrograde Cholangio-Pancreatography (ERCP) cannulation is wire guided. Up to now there is no doubt about the efficacy of such a procedure. The use of long wire requires the help of another person behind primary operator. The use of short wire rapid exchange allows the primary operator to perform all the steps by himself. Time of cannulation is known to be directly associated to post ERCP pancreatitis.

Aim of the study is to assess which length of guide wire allows the shorter cannulation time during primary ERCP. Post ERCP pancreatitis onset will be assessed for all patients

ELIGIBILITY:
Inclusion Criteria:

* indication to primary ERCP
* ASA (American Society of Anesthesiologists) 1, 2, 3

Exclusion Criteria:

* pancreas neoplasia
* pancreatitis
* ampulloma
* duodenum stenosis
* under mucous membrane haematoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2018-01-28 (Actual); Primary Completion 2018-01-28 (Actual); Study Completion 2025-12-14 (Estimated)

PRIMARY OUTCOMES:
Time of cannulation | 8 hours from intervention
  Time (in seconds) required to perform a complete and successful deep cannulation of the "biliary papilla" and the biliary tree assessed by timing it and reporting it in the prefashioned database

SECONDARY OUTCOMES:
Incidence of post ERCP pancreatitis | 8 hours post ERCP
  Incidence of post ERCP pancreatitis

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pugliese, MD, Study Chair — Niguarda Ca' Granda Hospital; Edoardo Forti, MD, Study Chair — Niguarda Ca' Granda Hospital; Raffaele Manta, MD, Study Chair — Niguarda Ca' Granda Hospital
Locations (1):
- Niguarda Hospital, Milan, Italy